CLINICAL TRIAL: NCT05680961
Title: Monitoring Movement Disorder Symptoms With a Mobile Medical App on Off-the-shelf Consumer Mobile Devices
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Parkinson's & Movement Disorders Center of Maryland (Other)
Collaborators: New Touch Digital Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NTD-101
Record Dates: First submitted 2022-06-21; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Parkinson's patients: Cohort of patients with clinical diagnosis of Parkinson's diseases with varied symptoms and severity.
  Interventions: Device: Monitoring Device

INTERVENTIONS:
Device: Monitoring Device — Monitoring Device

SUMMARY:
The purpose of this study is to evaluate whether New Touch Digital (NTD) NeuroRPM software installed on wearable devices can objectively measure and track symptoms in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subject is able to provide informed written consent
3. Subject has been clinically diagnosed with Parkinson's Disease
4. Subject is mentally and physically capable of performing tasks on the mobile device and related physical activities herein described

Exclusion Criteria:

1. Inability to give informed consent
2. Presence of additional neurological disease aside from the diseases being studied
3. Inability to understand and follow the directions for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is open to persons 18 years of age and older with a clinical diagnosis of Parkinson's diseases without other neurological diseases.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
NeuroRPM UPDRS predicted score vs. clinical raters' UPDRS | Comparison will be performed upon completion of the study, approximately in 1 year.
  We will compare symptom severity as predicted by NeuroRPM to UPDRS scores from clinical raters. Statistical significance will be evaluated by intraclass correlation and kappa-statistic.

CONTACTS AND LOCATIONS:
Locations (1):
- Parkinson's & Movement Disorders Center of Maryland, Elkridge, Maryland, United States

IPD SHARING:
Plan to Share IPD: No